CLINICAL TRIAL: NCT00433329
Title: COMPASS 3: An Open-label, Multi-Center Study Employing a Targeted 6-Minute Walk Test (6-MWT) Distance Threshold Approach to Guide Bosentan-Based Therapy and to Assess the Utility of Magnetic Resonance Imaging (MRI) on Cardiac Remodeling
Brief Title: Combination Therapy in Pulmonary Arterial Hypertension
Acronym: COMPASS 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-419
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; bosentan; sildenafil; combination therapy; Compass 3
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan; Sildenafil Citrate

ARMS (1):
- Bosentan (Experimental): Oral bosentan 62.5 mg twice daily (BID) first 4 weeks, followed by 24 weeks of 125 mg BID if the 62.5 mg BID dose was well tolerated, with the addition of sildenafil 20 mg thrice daily (TID) in patients who do not reach the 6-MWT distance threshold at Week 16
  Interventions: Drug: Bosentan; Drug: Sildenafil

INTERVENTIONS:
Drug: Bosentan — Oral bosentan 62.5 mg BID first 4 weeks followed by 24 weeks of 125 mg BID if the 62.5 mg BID dose was well tolerated
Drug: Sildenafil — Oral sildenafil 20 mg TID in patients who do not reach the 6-MWT distance threshold at Week 16

SUMMARY:
An open label, non-comparative study design is appropriate for this Phase 4 study designed to assess whether a core therapy of bosentan, either as monotherapy or with the addition of sildenafil, enables patients with pulmonary arterial hypertension (PAH) to achieve a 6-minute walk distance (6 MWD) of ≥380 meters after 28 weeks of therapy This design is also appropriate to pioneer the utility of cardiac MRI in assessing improved functional capacity in PAH and exploring its correlation with other parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-mandated procedures.
2. Males or females ≥ 12 years of age (females of child-bearing potential must have been surgically sterilized or use a reliable method of contraception).
3. Symptomatic patients with the following types of PAH belonging to World Health Organization (WHO) Pulmonary Hypertension Classification Group I:

   * Idiopathic (IPAH)
   * Familial (FPAH)
   * Associated with PAH (APAH):

     * Collagen vascular disease
     * Drugs and toxins
4. Patients naïve to treatment with advanced PAH therapies (i.e., endothelin receptor antagonists (ERAs), phosphodiesterase-5 (PDE-5) inhibitors or prostacyclins) with a right heart catheterization (RHC) showing all of the following:

   * Mean pulmonary arterial pressure (mPAP) ≥ 25 mm Hg
   * Pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg or left ventricular end diastolic pressure (LVEDP) ≤ 15 mm Hg when PCWP is not accurately obtained
   * Pulmonary vascular resistance ≥ 3 Wood units
5. 6-MWT distance ≥ 150 meters and < 360 meters.

Exclusion Criteria:

1. Patients with Pulmonary Hypertension (PH) belonging to WHO Classification Group II-V.
2. Patients with PAH (WHO PH Classification Group I) other than that listed in the Inclusion Criteria.
3. Pregnant and/or nursing.
4. Women of childbearing potential not using a reliable method of contraception.
5. Patients with known human immunodeficiency virus (HIV) infection.
6. Patients with significant vasoreactivity during right heart catheterization (i.e., a fall in mPAP to < 40 mm Hg with a decrease of ≥ 10 mm Hg and with a normal cardiac index ≥ 2.5 l/min.m^2).
7. Patients with restrictive lung disease (i.e., total lung capacity (TLC) < 60% of normal predicted value).
8. Patients with obstructive lung disease (i.e., forced expiratory volume/ forced vital capacity (FEV1/FVC) < 0.5).
9. Patients with impaired left ventricular function (LVEF <50%) or diastolic dysfunction.
10. Patients with portal hypertension, cirrhosis, moderate to severe liver impairment (Child-Pugh Class B or C), or liver enzymes (Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)) > 3.0 times the upper limit of normal range.
11. Treatment with glibenclamide (glyburide) and calcineurin inhibitors (cyclosporine A, tacrolimus) sirolimus, everolimus up to 1 week prior to Baseline (Day 1).
12. Patients currently receiving or predicted to require treatment, during the course of the study, with nitrates, protease inhibitors, or alpha-blockers.
13. Patients with a hemoglobin concentration < 75 % of the lower limit of the normal range or < 8.5 g/dL.
14. Patients currently receiving or predicted to require treatment with a prostanoid during the course of the study.
15. Patients with systolic blood pressure < 85 mm Hg.
16. Patients with body weight < 40 kg.
17. Patients who have received any investigational product within 90 days prior to Baseline.
18. Patients who previously received any advanced therapy for PAH (e.g., ERAs, PDE-5 inhibitors or prostacyclins).
19. Patients with hypersensitivity to sildenafil or any excipients of its formulation.
20. Patients with any contraindication to sildenafil treatment (i.e., nitrates).
21. Patients with any recent medical condition limiting the ability to comply with the study requirements (i.e., stroke, myocardial infarction).
22. Patients with unstable PAH whose disease state would prohibit the completion of study procedures, in the opinion of the investigator.
23. Patients unable to complete a MRI scan (e.g., claustrophobia).
24. Patients with permanent cardiac pacemakers, automatic internal cardioverter defibrillators (AICD's), neurostimulators, hearing aides, and other implanted metallic devices that are contraindicated during a MRI study.
25. Patients with conditions that would interfere with proper cardiac gating during MRI, such as atrial fibrillation or multiple premature ventricular contractions (PVCs)/premature atrial contractions (PACs).
26. Patients with conditions that prevent compliance with the protocol or the ability to adhere to therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

REFERENCES:
- [Derived] Benza RL, Raina A, Gupta H, Murali S, Burden A, Zastrow MS, Park MH, Simon MA. Bosentan-based, treat-to-target therapy in patients with pulmonary arterial hypertension: results from the COMPASS-3 study. Pulm Circ. 2018 Jan-Mar;8(1):2045893217741480. doi: 10.1177/2045893217741480. Epub 2017 Oct 24. PMID 29064349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 centers in the United States. First patient, first visit: 25 April 2007; last patient, last visit: 23 April 2010
Pre-assignment Details: The study included a screening phase of 2 weeks.
Groups:
- Bosentan/Sildenafil: Oral bosentan 62.5 mg twice daily (BID) for 4 week followed by 24 weeks of 125 mg BID with the addition of sildenafil 20 mg thrice daily (TID) in patients who do not reach the 6-MWT distance threshold at Week 16
Period: Overall Study
Arm/Group | Bosentan/Sildenafil
Started | 100
Completed | 79
Not Completed | 21
Not completed — Adverse Event | 9
Not completed — Death | 4
Not completed — Withdrew consent | 3
Not completed — Discontinued sildenafil | 2
Not completed — Moved out of state | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bosentan/Sildenafil
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (15.99)
Age, Customized [Number; unit: participants]
  Between 21 and 84 years | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reaching a 6-Minute Walk Test (6MWT) Distance ≥ 380 Meters
Description: The 6MWT is a non encouraged test, which measures the walking distance covered over a 6 minute period
Time Frame: at 16 weeks and at 28 weeks of a stepped approach to therapy
Population: Intention to treat population
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Bosentan/Sildenafil
Number analyzed (Participants) | 100
participants
  Week 16 | 16 [9.4 to 24.7]
  Week 28 | 24 [17.5 to 36.3]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected up to 24 hours after study drug discontinuation.
Arm/Group | Bosentan/Sildenafil
Serious Adverse Events (participants affected / at risk) | 30/100
Other Adverse Events (participants affected / at risk) | 88/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan/Sildenafil (N=100)
Anaemia (Blood and lymphatic system disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Death (General disorders) | 1
Generalised oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Malignant hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan/Sildenafil (N=100)
Anaemia (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 7
Oedema (General disorders) | 5
Oedema peripheral (General disorders) | 20
Bronchitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 6
Liver function test abnormal (Investigations) | 10
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No